CLINICAL TRIAL: NCT04785560
Title: Volumetrics and Proteomics in Shunted Normal Pressure Hydrocephalus
Acronym: LiNPH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Rafael T Holmgren, Principal investigator, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-00719
Record Dates: First submitted 2021-01-18; First posted 2021-03-08 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hydrocephalus, Normal Pressure; Ventriculomegaly, Cerebral; Shunt; Complications; Hydrocephalus Acquired
Keywords: Hydrocephalus, Normal Pressure; Ventriculomegaly, Cerebral; Shunt; Complications; Hydrocephalus Acquired; Volumetry; Proteomics; Cerebrospinal Fluid; Ventriculoperitoneal shunt; Synthetic MRI
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Shunt setting 4 (=110 mm H20) (Active Comparator): Patients randomised to have the Certas Plus valve initial shunt setting post-operatively set to 4 (110 mm H20), our standard setting.
  Interventions: Device: Initial shunt setting post-operatively of the Certas Plus shunt valve.
- Shunt setting 8 (=400 mm H20) (Active Comparator): Patients randomised to have the Certas Plus valve initial shunt setting post-operatively set to 8 (400 mm H20 a k a virtual off), in practice a closed non-functional shunt.
  Interventions: Device: Initial shunt setting post-operatively of the Certas Plus shunt valve.

INTERVENTIONS:
Device: Initial shunt setting post-operatively of the Certas Plus shunt valve. — The setting/resistance of the Certas Plus Shunt valve implanted is set according to randomisation and is not changed until the first post-operative MRI is performed 36-48 hours after surgery.
  Other Names: CODMAN CERTAS PLUS

SUMMARY:
Idiopathic normal pressure hydrocephalus (=iNPH) is a condition with disturbed circulation of cerebrospinal fluid (=CSF) causing symptoms such as balance and gait disorders, urinary incontinence and cognitive impairment in patients with cerebral ventricular dilation. The exact incidence is unknown but has been estimated at about 8.9% of the population over the age of 80 and the incidence is estimated to increase with an aging population. The symptoms can be temporarily improved by draining cerebrospinal fluid and so-called shunting (surgery with diversion of cerebrospinal fluid from the brain to the abdominal cavity). The symptoms and pathophysiology of iNPH are poorly described as well as the protein distribution in cerebrospinal fluid (proteomics) of the disease. There is also a need for improved diagnostical and prognostical tools that can guide in patient selection for surgery. The radiological tools in evaluating the disease and it´s progression need to be improved.

There is a shunt valve (Codman Certas Plus) used since 2015 that is widely used in clinical use and is well studied in research laboratories but little in clinical studies. The project aims to, before and after surgery, on patients with iNPH who will undergo investigation and shunting with Certas Plus at our department and in comparison with healthy controls: 1. Apply and evaluate a novel method to determine the volume of circulating CSF (volumetry). 2. Study the correlation between changes in volumetry and clinical outcome 3. Study NPH patients' distribution of proteins in cerebrospinal fluid and their change over time after shunting. 4. Evaluate the efficacy and functions of the Certas Plus valve.

In this way, the investigators hope to find increased knowledge about the NPH disease and its pathophysiology as well as useful instruments that can both predict the probability for a patient to be improved by a shunt operation and determine if a shunt has stopped working and thus be able to avoid unnecessary risky operations.

DETAILED DESCRIPTION:
BACKGROUND & SUMMARY DESCRIPTION OF THE PROJECT

Idiopathic normal pressure hydrocephalus (=iNPH) is a condition with disturbed cerebral dynamics causing symptoms in the form of balance and gait disorders, incontinence and cognitive impairment in patients with cerebral ventricular dilation. The condition is much more common than is generally known with a prevalence that increases sharply with age, from 2.1% in the age of 70 to 8.9% in ages over 80 years. Adams and Hakim described the disease as early as 1965 based on symptomatology and reversibility of symptoms after CSF tapping. However, it was not until 2005 that a compilation of evidence-based guidelines for the diagnosis and treatment of the disease came out, the iNPH International Guidelines. It was stated that at present, in addition to the CSF tap-test there is no reliable predictive test for a patient's likelihood to respond to shunting . There are several different scales for assessing the severity of the disease, one of which is the iNPH scale, with the subscales of gait, balance, neuropsychology and continence.

At the Department of Neurosurgery (NK) and Neurological (NL), Linköping University Hospital, there has been a well-functioning multi-professional team since 2004. The team investigates and treats iNPH with referrals coming from the Southeastern healthcare region of Sweden. Annually approximately 250 referrals are received, 70-80 patients are evaluated and at least 40 patients are operated with ventriculoperitoneal shunting. The evaluation consists in the first stage of radiological examinations, a clinical assessment by a neurologist, followed by motor assessment by a physiotherapist and cognitive assessment by an occupational therapist. CSF tap-tests are usually performed in which up to 50 ml of cerebrospinal fluid is drained by lumbar puncture, which in iNPH usually relieves the symptoms. Assessment also includes video recording of the movement pattern of a qualitative assessment. The results, together with the radiology, are weighed together and then the team if the patient should be offered treatment. The patients are operated with ventriculoperitoneal shunting at NK and followed up at NL with the same motor and cognitive tests three months after the operation, after which the results are evaluated. In larger studies, approximately 70 % of iNPH-patients receiving a shunt improve postoperatively.

Shunt therapy is the only treatment of iNPH and has been available since the 1950s. The goal of treatment is to reduce the amount of cerebrospinal fluid in the ventricular system and thereby normalize the volume in the ventricular system. Since the early 1990s adjustable shunt valves are increasingly used. This means that the valve if necessary can be adjusted after implantation with an external magnet applied to the site of the valve. The disadvantage of most adjustable valves is that the valve setting can be adjusted inadvertently when exposed to strong magnetic fields, for example if the patient undergoes a magnetic camera examination. Adjustable valves, however, bring many advantages as the resistance can be adapted to the patient's needs even after the operation. For example, one of the most common complications after shunting (subdural hematoma) can often be treated by raising the valve resistance. In 2015 the company Codman Johnson & Johnson introduced a novel shunt valve, Certas Plus, which is an adjustable shunt with eight different settings. The valve is established in clinical practice. Special features are the highest setting (8) which is 40 cm H20, which is a very high resistance which in theory should be equivalent to a turned off shunt and is called by the company "virtual off". It is also designed to be MR-resistant and thus does not change setting when exposed to a MRI magnetic field. These features have so far been tested in vitro but no clinical studies have yet been performed. The advantages of these functions are potentially fewer surgical procedures and inpatient care and also enables patients in the Southeastern healthcare region to carry out planned and acute MRI examinations in their home hospital without having to go to the Neurosurgical department in Linköping for valve readjustment.

Ventricular dilatation is a radiological diagnosis. Since the 1940s, the largest diameter between the lateral boundaries of the lateral ventricles and the largest biparietal diameter on the inside of the skull have been measured to obtain the so-called Evans index by dividing the two and obtaining the ratio. It is easy to measure but is a method with many sources of error and poor sensitivity to volume changes in the ventricular system. There is a need for a more reliable method in both clinical practice and research. Volumetry, i e measuring the volume of the ventricles, has become an increasingly used method which, however, has not yet taken place in clinical practice due to time-consuming manual calculation. With MRI images that are converted in a special software (ITK-SNAP), the volume may be calculated and a three-dimensional image of the ventricular system can be plotted. A few studies in the literature have studied the relationship between shunt valves resistance and reduction in ventricular volume. There are no prospective blinded studies studying the change in ventricular volume related to shunt therapy, shunt resistance, nor are there any studies on whether there is a correlation between ventricular volume reduction and postoperative clinical outcome. A study group in Uppsala has recently published a study on shunted iNPH-patients where a novel MRI-technology developed in Linköping (SyntheticMR) clearly can show how ventricular volume decreases after treatment without changing Evans' index. In the same study, it was also possible to show how another parameter in the ventricles, the so-called callosal angle, clearly changes after shunting. This is part of a radiological assessment scale, Radscale, which can be applied to this patient group. The same research group has previously also been able to show with SyntheticMR how the ventricular volume decreases after tap tests on iNPH patients to be restored to the original within 24 hours. CMIV (=Center for Medical Imaging and Visualization) at US Linköping has several of the University Hospital's 3-Tesla MR cameras and a good technological and scientific knowledge of SyntheticMR as the method is developed there. Using a short MRI protocol (6 minutes), it produces quantitative data of the condition of the brain tissue, which makes it easy to ascertain what is gray and white brain matter, the brain cells' support protein myelin as well as cerebrospinal fluid and calculates the volume of each component. Sequences with standard protocols for hydrocephalus, including DTI (=Diffusion Tensor Imaging) sequences, require an additional 15-20 minutes in the MRI camera. SyntheticMR can also as the hitherto only method easily calculate the volume of CSF that is located outside of the ventricles in the basal cisterns and brain sulci. However, no one has so far studied the volumes of extracerebral CSF in the healthy brain or in iNPH. In addition, no one has studied how this volume extracerebral CSF changes in response to shunting.

The proteome is the collective name of the proteins that an organism or an organ synthesizes. The proteome is not constant but varies between different organs in the same organism and in the same organ over time and change in the diseased organism or organ. Proteomics is the science of these proteins and can be used to examine when and where certain proteins can be found, concentrations of these, how they are broken down, modified and interact in various physiological and disease processes. Some neurological diseases have been characterized in their proteomic alterations, such as essential tremor and chronic neuropathic pain, by the members of our for research group. The proteomics of the cerebrospinal fluid in patients with iNPH is relatively unexplored with only three studies in the literature. These have characterized a few proteins that stand out compared to what is expected in a healthy brain. No comparative studies between CSF taken via lumbar puncture and cerebrospinal fluid from the ventricles have been performed. At the department of Pain- and Rehabilitational medicine at Linköping University Hospital a proteomics lab (PAINOMICS lab) with many scientific publications is established. The standard methods available for proteomics studies are two-dimensional gel electrophoresis (2D electrophoresis) and mass spectrometry (LC-MS/MS). These are applied to analyze up to a thousand proteins in one sample and with antibody-based technology validate them. With antibody-based technology, one can also analyze up to 86 cytokines, chemokines, growth factors and metabolic substances in a so-called multiplex panel. The data sets obtained in proteomic studies are complex. These datasets are made up of many and highly correlated variables (concentrations of proteins). One can then compare content changes of proteins between patients with iNPH and controls establish a difference in "fingerprint" of the proteome. There is a great need for new biomarkers as a complement to currently available methods for making a definite diagnosis, assessing the probability that the therapy will be successful and creating a deeper understanding of the pathophysiology of iNPH.

OBJECTIVES, SCIENTIFIC ISSUES AND SUBSTUDIES:

1. Evaluate and validate a clinically useful method of monitoring ventricular volumes with Synthetic MRI. Comparison against an established volumetric method (ITK-SNAP) and for intra- and inter-assessor reliability.
2. Map ventricular volumes and amount extracerebral intracranial CSF during normal physiological conditions in healthy control persons and of INPH patients and calculate how these volumes change after shunting in INPH.
3. Investigate how volume change and change in volumetry and iNPH Radscale after shunting correlate to clinical outcome 3 months postoperatively.
4. Examine the shunt valve CERTAS PLUS for its function and safety for MR resistance in vivo and correlate the degree of reduction in ventricular volume based on the resistance of the valve.
5. Map the proteomic expression of iNPH in CSF and blood plasma pre-operatively and monitor change at 3, 12 and 36 months after ventriculoperitoneal shunting.
6. Compare how the proteomics in CSF in iNPH differ between lumbar and ventricular CSF and blood plasma. Examine whether the iNPH patients lumbar CSF is different compared to a neurologically healthy cohort control persons of similar age and patients with essential tremor.

PROJECT PLAN, IMPLEMENTATION AND SELECTION OF RESEARCH OBJECTS:

The Swedish National Ethics Review board (Etikprövningsmyndigheten), ref no 2020-0071920, has approved this project plan.

Fifty patients who have undergone the NPH team's investigation and are deemed suitable for shunt treatment are recruited consecutively for the study.

A control group consisting of 50 volunteer individuals over 60 years of age is recruited via the operation waiting list of the departments of Orthopedics, Urology and Gynaecology at Linköping University Hospital. Volunteers will be recruited from elderly patients who during planned orthopedic/gynecological/urological surgery in spinal anesthesia will undergo a lumbar puncture for the application of the anesthesia. Volunteers will preoperatively undergo an MRI examination including standard sequences as well as SyntheticMR protocols for volumetry.

The NPH team's pre-operative investigation of iNPH patients consists of the following examinations: 1. Clinical assessment by a neurologist. 2. Balance and ability to walk is assessed by a physiotherapist. Tests include Timed Up and Go (TUG) , number of steps and time as well as gait scale, balance scale and 10 m walking as part of the iNPH scale. 3. An occupational therapist assesses the cognitive functions and performs the following tests: MMSE (=Mini-Mental State Examination), Grooved pegboard, Rey Auditory Verbal Learning Test, Stroop color naming and Stroop interference , Trail Making Test A and B. 4. Estimation of urinary incontinence is done on the urinary incontinence scale. All assessments are combined in the iNPH scale.

A lumbar puncture with measuring of intrathecal pressure, analysis of cells, protein, antibodies against Lyme disease and the CSF tap-test is included in the basic investigation. The patient's medical history, symptoms and results from radiology and CSF tap-test are discussed within the NPH team to decide whether the patient is deemed suitable for a shunt.

Patients who are recommended shunting by the team and do not meet the study's exclusion criteria are called to a outpatients visit to Dr Rafael Holmgren, are informed of the intended operation and associated risks and offered study participation after oral and written information. Patients are offered time to think and get back to the contact nurse's telephone before answering.

Volunteers in the control group are recruited among patients planned for surgery in spinal anestesia by the departments of Orthopedics, Urology and Gynaecology at Linköping University Hospital. They are informed of possible participation in the study orally by telephone or if so desired during an outpatient consultation with Dr Rafael Holmgren in addition to written information. Participants in the control group will before their operation undergo an MRI-examination with standard protocol and Synthetic MRI. Before spinal anaesthesia is administered 10 ml of lumbar CSF is drawn for analysis of the proteomic profile as is a blood sample for the same purpose.

Participating iNPH-patients to be shunted will the day before the surgery undergo an MRI with modified standard protocol and SyntheticMR; time required is about 45 minutes.

The patients undergo general anesthesia the following day and a lumbar puncture is performed, after which 10 ml of cerebrospinal fluid is collected. Simultaneously, a blood sample is also taken for proteomic analysis. The patient is operated with ventriculoperitoneal shunting by a standard procedure by one of three surgeons (Dr Rafael Holmgren, Dr Peter Zsigmond or Dr Martin Nilsson at NK). Patients receive a Codman CERTAS PLUS shunt valve with one out of two valve settings blinded to the operator, patient and radiological investigators (set by another colleague in accordance with randomization): 4 (=110 mm H20 , conventional default setting) or 8 (>400 mm H20 a k a "virtual off"). As the cerebral ventricles are punctured by the catheter another 10 ml CSF for proteomics is collected here. The samples are transported to the proteomics laboratory, centrifuged, aliquoted into small aliquots before being frozen. They are then stored in the biobank at Occupational and Environmental Medicine at the Linköping University Hospital (registered with the National Board of Health and Welfare). Each incoming subject is given a unique code number and all test tubes are marked with this number. The code key is kept in a locked cabinet at the Department of Neurosurgery in Linköping.

Approximately 36 hours (range 24-48 hours) after the operation, the patient undergoes a new MRI examination with SyntheticMR and after this examination, the valve setting is checked with a reader compass held over the valve. The patients who initially received setting 8 of the valve are now adjusted to receive the standard setting 4, unless they have suffered a subdural hematoma after the operation, which is detected in the MRI examination postoperatively. The patient is then discharged to either the home or their local hospital. Thus, all patients return home with a functioning shunt treatment.

The patients are called back for standard follow-up for shunted iNPH patients after three months for a return visit to the surgeon and carry out a clinical examination/follow-up by a physiotherapist and occupational therapist with the same protocol for the motor and cognitive tests as before the operation. Patients also undergo a new MRI examination with the same protocol as before the operation. The shunt valve setting is checked after the MRI to confirm that the valve setting is the same as before. Also, the shunt valve chamber is punctured under sterile conditions with a small needle to obtain 10 ml of CSF from the ventricles and a blood sample is also taken for proteomic analysis.

Patients are called back to the operating physician one and three years after the operation for clinical assessment and new puncture of the shunt valve and blood tests with the same procedure as at the 3-month check-up.

All shunt-related complications, including adjustments of the shunt resistance in connection with MRI, are registered continuously.

CSF- and blood samples assays are performed by Professor Bijar Ghafouri at Painomics lab with both mass spectrometry and 2D-electrophoresis to identify, separate the proteins and ELISA techniques to characterize them. The identity of the sample is blinded to the examiner.

MRI studies are analyzed in a specific software adapted for assessment of volumes in studies made with both conventional technology (ITK SNAP) and SyntheticMR technology by Dr Holmgren and Dr. Georgiopoulos. The patient's identity and shunt setting are blinded to the examiners as well as timing of the study.

STATISTICAL BASIS FOR THE SIZE OF THE STUDY POPULATION

An amount of fifty iNPH-patients is judged adequate to answer the project's stated objectives. This is because the studies in proteomics at iNPH (by Chen et al and Li et al, see references) included 18 and 15 patients, respectively, and obtained clear statistically significant results. The studies on ventricular volume calculated with Synthetic MRI after lumbar puncture and shunting by Virhammar et al included 23 and 18 patients, respectively, and gave clear statistically significant results. The number of neurologically healthy control subjects/volunteers in the control group amounts to 50 to correspond to the number INPH patients.

ELIGIBILITY:
FOR iNPH-PATIENTS:

INCLUSION CRITERIA:

* Must meet the clinical criteria for iNPH according to the International Guide lines of 2005
* Must undergo shunt implantation at the Dpt of Neurosurgery Linköping University Hospital.

EXCLUSION CRITERIA:

* Individuals not able to participate/cooperate in study tasks with regard to cognitive symptoms
* Individuals with claustrophobia that makes awake MRI examination impossible.
* Individuals with implants that make MRI examination impossible (for instance pacemaker, refers only to the MRI examinations included in the study).
* Patients with severe co-existing chronical neurological diseases (refers only to the proteomic examinations included in the study).

FOR CONTROL GROUP VOLUNTEERS:

INCLUSION CRITERIA:

* Must undergo surgery under spinal anesthesia at the Dpt of Orthopaedics, Urology or Gynaecology at the University Hospital Linkoping.
* Must consider themselves neurologically healthy and have not undergone neurological disease.

EXCLUSION CRITERIA:

* Individuals with claustrophobia that makes awake MRI examination impossible.
* Individuals with implants that make MRI examination impossible
* Individuals with malignant disease or oncological treatment for such disease.
* Individuals with neurological disorders detected after study MRI.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in Idiopathic normal pressure hydrocephalus scale | Assessed within 3 months pre-operatively and 3 months post-operatively.
  A validated, continuous, calibrated and norm-based scale for the grading of severity and assessment of treatment outcome in idiopathic normal pressure hydrocephalus (iNPH). Designed for the assessment of the four domains, gait, neuropsychology, balance and continence, using ordinal ratings and continuous measures. A value of 100 represents normal function and 0 the most severe level of dysfunction.
Change from baseline CSF volume at 2 days postoperatively. | Assessed on MRI scan 36-48 hours post-operatively.
  Volume of the CSF contained 1. in the cerebral ventricular system. 2. Intracranially outside the cerebral ventricular system. Measured by means of Synthetic MRI. Baseline values are collected at the MRI-scan the day before surgery.
Change from baseline CSF volume at 3 months post-operatively. | Assessed on MRI scan 3 months post-operatively
  Volume of the CSF contained 1. in the cerebral ventricular system. 2. Intracranially outside the cerebral ventricular system. Measured by means of Synthetic MRI. Baseline values are collected at the MRI-scan the day before surgery.
Change from Baseline iNPH Radscale at 2 Days post-operatively. | Assessed on MRI scan 36-48 hours post-operatively and 3. 3 months post-operatively
  A radiological scale to standardize the evaluation of radiological morphological signs in iNPH. Ranging from 0 to 12, a high iNPH Radscale score combined with clinical symptoms should raise suspicion of iNPH. Baseline value is aquired at the MRI-scan the day before surgery.
Change from Baseline iNPH Radscale at 3 months post-operatively. | Assessed on MRI scan 3 months post-operatively.
  A radiological scale to standardize the evaluation of radiological morphological signs in iNPH. Ranging from 0 to 12, a high iNPH Radscale score combined with clinical symptoms should raise suspicion of iNPH. Baseline value is aquired at the MRI-scan the day before surgery.
Number of participants with shunt complications | From the day of surgery until 3 months post-operatively.
  Complications are defined as adverse effects of shunt surgery such as misplacement, dislocation, obstruction, malfunction, post-operative bleeding (subdural hematoma) and shunt infection.
Proteomic pattern of alpha-1B-glycoprotein in lumbar, ventricular CSF and blood plasma. | Assessed from intra-operative samples the day of surgery, 3-, 12- and 36-months post-operatively.
  The proteome is the entire set of proteins that is produced or modified by an organism or organ system. Proteomics generally refers to the large-scale experimental analysis of proteins and proteomes, in this case the iNPH disease specific pattern of proteins present in the above mentioned body fluids where the concentration of multiple proteins can be elevated or lowered compared with healthy subjects.
  More specifically we will study the concentration of alpha-1B-glycoprotein compared with healthy subjects, change of concentration compared to baseline at 3-, 12- and 36-months post-operatively.
Proteomic pattern of apolipoproteins A-1 & A-IV in lumbar, ventricular CSF and blood plasma. | Assessed from intra-operative samples the day of surgery, 3-, 12- and 36-months post-operatively.
  The proteome is the entire set of proteins that is produced or modified by an organism or organ system. Proteomics generally refers to the large-scale experimental analysis of proteins and proteomes, in this case the iNPH disease specific pattern of proteins present in the above mentioned body fluids where the concentration of multiple proteins can be elevated or lowered compared with healthy subjects.
  More specifically we will study the concentration of apolipoproteins A-1 & A-IV compared with healthy subjects, change of concentration compared to baseline at 3-, 12- and 36-months post-operatively.
Proteomic pattern of alpha-1-antitrypsin in lumbar, ventricular CSF and blood plasma. | Assessed from intra-operative samples the day of surgery, 3-, 12- and 36-months post-operatively.
  The proteome is the entire set of proteins that is produced or modified by an organism or organ system. Proteomics generally refers to the large-scale experimental analysis of proteins and proteomes, in this case the iNPH disease specific pattern of proteins present in the above mentioned body fluids where the concentration of multiple proteins can be elevated or lowered compared with healthy subjects.
  More specifically we will study the concentration of alpha-1-antitrypsin compared with healthy subjects, change of concentration compared to baseline at 3-, 12- and 36-months post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zsigmond, MD, ass prof, Study Director — Assistant professor
Locations (1):
- Neurosurgical department University Hospital Linköping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams RD, Fisher CM, Hakim S, Ojemann RG, Sweet WH. SYMPTOMATIC OCCULT HYDROCEPHALUS WITH "NORMAL" CEREBROSPINAL-FLUID PRESSURE. A TREATABLE SYNDROME. N Engl J Med. 1965 Jul 15;273:117-26. doi: 10.1056/NEJM196507152730301. No abstract available. PMID 14303656
- [Background] Marmarou A, Bergsneider M, Klinge P, Relkin N, Black PM. The value of supplemental prognostic tests for the preoperative assessment of idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Sep;57(3 Suppl):S17-28; discussion ii-v. doi: 10.1227/01.neu.0000168184.01002.60. PMID 16160426
- [Background] Marmarou A, Bergsneider M, Relkin N, Klinge P, Black PM. Development of guidelines for idiopathic normal-pressure hydrocephalus: introduction. Neurosurgery. 2005 Sep;57(3 Suppl):S1-3; discussion ii-v. doi: 10.1227/01.neu.0000168188.25559.0e. PMID 16160424
- [Background] Toma AK, Papadopoulos MC, Stapleton S, Kitchen ND, Watkins LD. Systematic review of the outcome of shunt surgery in idiopathic normal-pressure hydrocephalus. Acta Neurochir (Wien). 2013 Oct;155(10):1977-80. doi: 10.1007/s00701-013-1835-5. Epub 2013 Aug 23. PMID 23975646
- [Background] Shellock FG, Bedwinek A, Oliver-Allen M, Wilson SF. Assessment of MRI issues for a 3-T "immune" programmable CSF shunt valve. AJR Am J Roentgenol. 2011 Jul;197(1):202-7. doi: 10.2214/AJR.10.5915. PMID 21701031
- [Background] Bergsneider M, Black PM, Klinge P, Marmarou A, Relkin N. Surgical management of idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Sep;57(3 Suppl):S29-39; discussion ii-v. doi: 10.1227/01.neu.0000168186.45363.4d. PMID 16160427
- [Background] Czosnyka Z, Pickard JD, Czosnyka M. Hydrodynamic properties of the Certas hydrocephalus shunt. J Neurosurg Pediatr. 2013 Feb;11(2):198-204. doi: 10.3171/2012.10.PEDS12239. Epub 2012 Dec 7. PMID 23215818
- [Background] Kockum K, Lilja-Lund O, Larsson EM, Rosell M, Soderstrom L, Virhammar J, Laurell K. The idiopathic normal-pressure hydrocephalus Radscale: a radiological scale for structured evaluation. Eur J Neurol. 2018 Mar;25(3):569-576. doi: 10.1111/ene.13555. Epub 2018 Feb 2. PMID 29281156
- [Background] Leinonen V, Koivisto AM, Savolainen S, Rummukainen J, Sutela A, Vanninen R, Jaaskelainen JE, Soininen H, Alafuzoff I. Post-mortem findings in 10 patients with presumed normal-pressure hydrocephalus and review of the literature. Neuropathol Appl Neurobiol. 2012 Feb;38(1):72-86. doi: 10.1111/j.1365-2990.2011.01195.x. PMID 21696417
- [Background] Ambarki K, Israelsson H, Wahlin A, Birgander R, Eklund A, Malm J. Brain ventricular size in healthy elderly: comparison between Evans index and volume measurement. Neurosurgery. 2010 Jul;67(1):94-9; discussion 99. doi: 10.1227/01.NEU.0000370939.30003.D1. PMID 20559096
- [Background] Toma AK, Holl E, Kitchen ND, Watkins LD. Evans' index revisited: the need for an alternative in normal pressure hydrocephalus. Neurosurgery. 2011 Apr;68(4):939-44. doi: 10.1227/NEU.0b013e318208f5e0. PMID 21221031
- [Background] McConnell KA, Zou KH, Chabrerie AV, Bailey NO, Black PM. Decreases in ventricular volume correlate with decreases in ventricular pressure in idiopathic normal pressure hydrocephalus patients who experienced clinical improvement after implantation with adjustable valve shunts. Neurosurgery. 2004 Sep;55(3):582-92; discussion 592-3. doi: 10.1227/01.neu.0000134385.23401.01. PMID 15335425
- [Background] Virhammar J, Laurell K, Cesarini KG, Larsson EM. Increase in callosal angle and decrease in ventricular volume after shunt surgery in patients with idiopathic normal pressure hydrocephalus. J Neurosurg. 2019 Jan 1;130(1):130-135. doi: 10.3171/2017.8.JNS17547. Epub 2018 Feb 2. PMID 29393749
- [Background] Virhammar J, Warntjes M, Laurell K, Larsson EM. Quantitative MRI for Rapid and User-Independent Monitoring of Intracranial CSF Volume in Hydrocephalus. AJNR Am J Neuroradiol. 2016 May;37(5):797-801. doi: 10.3174/ajnr.A4627. Epub 2015 Dec 24. PMID 26705322
- [Background] West J, Warntjes JB, Lundberg P. Novel whole brain segmentation and volume estimation using quantitative MRI. Eur Radiol. 2012 May;22(5):998-1007. doi: 10.1007/s00330-011-2336-7. Epub 2011 Nov 24. PMID 22113264
- [Background] Zsigmond P, Ljunggren SA, Ghafouri B. Proteomic Analysis of the Cerebrospinal Fluid in Patients With Essential Tremor Before and After Deep Brain Stimulation Surgery: A Pilot Study. Neuromodulation. 2020 Jun;23(4):502-508. doi: 10.1111/ner.13075. Epub 2019 Nov 22. PMID 31755628
- [Background] Olausson P, Ghafouri B, Backryd E, Gerdle B. Clear differences in cerebrospinal fluid proteome between women with chronic widespread pain and healthy women - a multivariate explorative cross-sectional study. J Pain Res. 2017 Mar 13;10:575-590. doi: 10.2147/JPR.S125667. eCollection 2017. PMID 28331360
- [Background] Chen CPC, Huang YC, Chang CN, Chen JL, Hsu CC, Lin WY. Changes of cerebrospinal fluid protein concentrations and gait patterns in geriatric normal pressure hydrocephalus patients after ventriculoperitoneal shunting surgery. Exp Gerontol. 2018 Jun;106:109-115. doi: 10.1016/j.exger.2018.01.027. Epub 2018 Feb 2. PMID 29408782
- [Background] Li X, Miyajima M, Mineki R, Taka H, Murayama K, Arai H. Analysis of potential diagnostic biomarkers in cerebrospinal fluid of idiopathic normal pressure hydrocephalus by proteomics. Acta Neurochir (Wien). 2006 Aug;148(8):859-64; discussion 864. doi: 10.1007/s00701-006-0787-4. Epub 2006 Jun 6. PMID 16755327
- [Background] Yushkevich PA, Yang Gao, Gerig G. ITK-SNAP: An interactive tool for semi-automatic segmentation of multi-modality biomedical images. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:3342-3345. doi: 10.1109/EMBC.2016.7591443. PMID 28269019
- [Background] Hellstrom P, Klinge P, Tans J, Wikkelso C. A new scale for assessment of severity and outcome in iNPH. Acta Neurol Scand. 2012 Oct;126(4):229-37. doi: 10.1111/j.1600-0404.2012.01677.x. Epub 2012 May 16. PMID 22587624
- [Background] Scollato A, Terreni A, Caldini A, Salvadori B, Gallina P, Francese S, Mastrobuoni G, Pieraccini G, Moneti G, Bini L, Messeri G, Di Lorenzo N. CSF proteomic analysis in patients with normal pressure hydrocephalus selected for the shunt: CSF biomarkers of response to surgical treatment. Neurol Sci. 2010 Jun;31(3):283-91. doi: 10.1007/s10072-009-0181-0. Epub 2009 Nov 21. PMID 19936883
- [Result] Andersson J, Rosell M, Kockum K, Lilja-Lund O, Soderstrom L, Laurell K. Prevalence of idiopathic normal pressure hydrocephalus: A prospective, population-based study. PLoS One. 2019 May 29;14(5):e0217705. doi: 10.1371/journal.pone.0217705. eCollection 2019. PMID 31141553